CLINICAL TRIAL: NCT05614986
Title: Prospective Evaluation of Neurocognition in Patients Undergoing Transcatheter Aortic Valve Replacement: Periprocedural Changes and Predictors of Improvement
Brief Title: Prospective Evaluation of Neurocognition in Patients Undergoing Transcatheter Aortic Valve Replacement
Acronym: Neurcog TAVR
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 021-262
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Aortic Stenosis
Keywords: TAVR; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Cognitive Dysfunction; Aortic Valve Stenosis | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Mild Cognitive Impairment Undergoing TAVR: Patients will be treated with standard of care. In addition, patients will complete the mini MoCA at 3 time points
  Interventions: Other: 5 minute Montreal Cognitive Assessment (mini MoCA)

INTERVENTIONS:
Other: 5 minute Montreal Cognitive Assessment (mini MoCA) — The mini MoCA will be completed by the patient before TAVR, and 30 days and 6 months after TAVR

SUMMARY:
This trail is for patients with mild cognitive impairment (MCI) who are receiving a transcatheter aortic valve replacement (TAVR). We will assess changes in neurocognition following TAVR with the 5 minute Montreal Cognitive Assessment (mini MoCA) when comparing pre procedure with post procedure assessments.

DETAILED DESCRIPTION:
Patients with mild cognitive impairment who are being treated with a TAVR can choose to take part in this trial. This trial will prospectively enroll patients at 4 Baylor Scott & White facilities. 80 patients will be enrolled between all sites. The mini MoCA will be conducted at the following time points: pre TAVR, 30 days post TAVR, and 6 months post TAVR. All other data will be collected from patient charts and are considered standard part of their care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Undergoing a TAVR procedure
3. Possible MCI as determined by procedures already used in the TAVR clinics, including 1 of the 4:

   1. MMSE < 27
   2. History of MCI, dementia, or stroke (CVA or TIA)
   3. History of prescription treatment for MCI
   4. Discretion of the investigator, physician, or clinic staff
4. Scores 25 or less on the mini MoCA exam

Exclusion Criteria:

1. In another research study that doesn't allow dual enrolment, or dual enrolment has not been granted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TAVR with mild cognitive impairment
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Neurocognition measured by Mini MoCA at 30 days post TAVR | 30 days post TAVR
  Changes in neurocognition compared to baseline at 30 days

SECONDARY OUTCOMES:
Neurocognition measured by Mini MoCA at 6 months post TAVR | 6 months post TAVR
  Changes in neurocognition compared to baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasa Potluri, MD, Principal Investigator — Baylor Scott and White The Heart Hospital Plano
Locations (4):
- United States (4):
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Baylor Scott & White All Saints at Fort Worth, Fort Worth, Texas
  - Baylor Scott and White The Heart Hospital Baylor Plano, Plano, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Result] Auffret V, Campelo-Parada F, Regueiro A, Del Trigo M, Chiche O, Chamandi C, Allende R, Cordoba-Soriano JG, Paradis JM, De Larochelliere R, Doyle D, Dumont E, Mohammadi S, Cote M, Marrero A, Puri R, Rodes-Cabau J. Serial Changes in Cognitive Function Following Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2016 Nov 15;68(20):2129-2141. doi: 10.1016/j.jacc.2016.08.046. Epub 2016 Sep 28. PMID 27692728
- [Result] Potluri S, Szerlip M, Al-Azizi K, Harrington K, Kodali S, Kapadia S, Lu M, Leon MB, Mack MJ. Neurocognitive Function Change in Low-Risk Patients Undergoing TAVR Versus SAVR: Insights From PARTNER-3. JACC Cardiovasc Interv. 2020 Nov 23;13(22):2713-2714. doi: 10.1016/j.jcin.2020.08.009. No abstract available. PMID 33213758
- [Result] Arevalo-Rodriguez I, Smailagic N, Roque I Figuls M, Ciapponi A, Sanchez-Perez E, Giannakou A, Pedraza OL, Bonfill Cosp X, Cullum S. Mini-Mental State Examination (MMSE) for the detection of Alzheimer's disease and other dementias in people with mild cognitive impairment (MCI). Cochrane Database Syst Rev. 2015 Mar 5;2015(3):CD010783. doi: 10.1002/14651858.CD010783.pub2. PMID 25740785
- [Result] O'Bryant SE, Humphreys JD, Smith GE, Ivnik RJ, Graff-Radford NR, Petersen RC, Lucas JA. Detecting dementia with the mini-mental state examination in highly educated individuals. Arch Neurol. 2008 Jul;65(7):963-7. doi: 10.1001/archneur.65.7.963. PMID 18625866
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Khan MM, Herrmann N, Gallagher D, Gandell D, Fremes SE, Wijeysundera HC, Radhakrishnan S, Sun YR, Lanctot KL. Cognitive Outcomes After Transcatheter Aortic Valve Implantation: A Metaanalysis. J Am Geriatr Soc. 2018 Feb;66(2):254-262. doi: 10.1111/jgs.15123. Epub 2017 Nov 21. PMID 29159840
- [Result] Liew TM. The Optimal Short Version of Montreal Cognitive Assessment in Diagnosing Mild Cognitive Impairment and Dementia. J Am Med Dir Assoc. 2019 Aug;20(8):1055.e1-1055.e8. doi: 10.1016/j.jamda.2019.02.004. Epub 2019 Mar 23. PMID 30910550
- [Result] Wong A, Nyenhuis D, Black SE, Law LS, Lo ES, Kwan PW, Au L, Chan AY, Wong LK, Nasreddine Z, Mok V. Montreal Cognitive Assessment 5-minute protocol is a brief, valid, reliable, and feasible cognitive screen for telephone administration. Stroke. 2015 Apr;46(4):1059-64. doi: 10.1161/STROKEAHA.114.007253. Epub 2015 Feb 19. PMID 25700290
- [Result] Roalf DR, Moore TM, Wolk DA, Arnold SE, Mechanic-Hamilton D, Rick J, Kabadi S, Ruparel K, Chen-Plotkin AS, Chahine LM, Dahodwala NA, Duda JE, Weintraub DA, Moberg PJ. Defining and validating a short form Montreal Cognitive Assessment (s-MoCA) for use in neurodegenerative disease. J Neurol Neurosurg Psychiatry. 2016 Dec;87(12):1303-1310. doi: 10.1136/jnnp-2015-312723. Epub 2016 Apr 12. PMID 27071646
- See also: MoCA Cognitive Assessment — https://www.mocatest.org/paper/